CLINICAL TRIAL: NCT03031652
Title: Clinical Analysis of Ocular Parameters Contributing to Intraoperative Pain During Standard Phacoemulsification
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Hong Kyun Kim, M.D, Professor, Kyungpook National University Hospital
Other Study IDs: KNUH
Record Dates: First submitted 2017-01-20; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Phacoemulsification
Keywords: pain; axial length; anterior chamber depth; intraocular pressure
MeSH Terms: conditions — Pain | interventions — Phacoemulsification

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled group: Patients who had senile cataract and underwent phacoemulsification with topical anesthesia.
  Interventions: Device: Phacoemulsification

INTERVENTIONS:
Device: Phacoemulsification — The device device used to provide and perform small profile entry for cataract extraction with or without option of insertion of a specified intraocular lens implant
  Other Names: INFINITI® Vision System

SUMMARY:
Charts of 142 patients who underwent standard phacoemulsification under topical anesthesia between March and August 2016 were reviewed. The pain during phacoemulsification and 1 h after surgery was assessed and compared using a visual analog scale.

DETAILED DESCRIPTION:
Patients scheduled for elective phacoemulsification and intraocular lens implantation with the Infiniti Vision System (Alcon, Fort Worth, USA) were included. All operations were performed in Kyungpook National University Hospital by the same surgeon between March and August 2016.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent phacoemulsification with topical anesthesia

Exclusion Criteria:

* Patients who needed general anesthesia or were taking medications capable of affecting perceived pain
* Patients who had traumatic cataract and/or conditions likely to require vitrectomy and trans-scleral fixation of posterior chamber intraocular lens

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had senile cataract and needed to receive cataract surgery (phacoemulsification) under topical anesthesia were included.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Pain score assessed with Visual Analogue Scale (VAS) | 1 hour after the end of surgery
  Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
  A third person assessed subjective pain using a pain visual analog scale ranging from 0 (no pain) to 10 (worst pain imaginable) after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Kyun Kim, M.D.,Ph.D., Study Director — Department of ophthalmology, Kyungpook national university hospital
Locations (1):
- Kyungpook national university hospital, Daegu, Samduk-2ga, Jung-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fichman RA. Use of topical anesthesia alone in cataract surgery. J Cataract Refract Surg. 1996 Jun;22(5):612-4. doi: 10.1016/s0886-3350(96)80019-8. PMID 8784636
- [Background] O'Brien PD, Fulcher T, Wallace D, Power W. Patient pain during different stages of phacoemulsification using topical anesthesia. J Cataract Refract Surg. 2001 Jun;27(6):880-3. doi: 10.1016/s0886-3350(00)00757-4. PMID 11408135
- [Background] Ursea R, Feng MT, Zhou M, Lien V, Loeb R. Pain perception in sequential cataract surgery: comparison of first and second procedures. J Cataract Refract Surg. 2011 Jun;37(6):1009-14. doi: 10.1016/j.jcrs.2011.01.020. PMID 21596244
- [Background] Cho YK, Chang HS, Kim MS. Risk factors for endothelial cell loss after phacoemulsification: comparison in different anterior chamber depth groups. Korean J Ophthalmol. 2010 Feb;24(1):10-5. doi: 10.3341/kjo.2010.24.1.10. Epub 2010 Feb 5. PMID 20157408
- [Background] Zauberman H. Extreme deepening of the anterior chamber during phacoemulsification. Ophthalmic Surg. 1992 Aug;23(8):555-6. PMID 1508488
- [Background] Ezra DG, Allan BD. Topical anaesthesia alone versus topical anaesthesia with intracameral lidocaine for phacoemulsification. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD005276. doi: 10.1002/14651858.CD005276.pub2. PMID 17636793
- [Result] Nahra Saad D, Castilla Cespedes M, Martinez Palmer A, Pazos Lopez M. Phacoemulsification and lens-iris diaphragm retropulsion syndrome. Ophthalmic Surg Lasers Imaging. 2005 Nov-Dec;36(6):512-3. PMID 16355958